CLINICAL TRIAL: NCT02916498
Title: Field Shape and Amplitude Sensitivity Exploratory Study (CONTOUR Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to a business decision
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A4062
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Neuropathic Pain in the Low Back and Legs
Keywords: chronic neuropathic pain in the low back and legs; subperception spinal cord stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bipolar then alternative field shape stimulation (Active Comparator): Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System: Spinal cord stimulation for the management of chronic neuropathic pain programmed with bipolar stimulation for 21 days, then alternative field shape stimulation for 21 days
  Interventions: Device: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System
- Alternative then bipolar field shape stimulation (Experimental): Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System: Spinal cord stimulation for the management of chronic neuropathic pain programmed with alternative field shape stimulation for 21 days, then bipolar stimulation for 21 days
  Interventions: Device: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System

INTERVENTIONS:
Device: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System — Spinal cord stimulation for the management of chronic neuropathic pain

SUMMARY:
The study aims to better understand how to program Spinal Cord Stimulation for the treatment of chronic low back and leg pain

ELIGIBILITY:
Key Inclusion Criteria:

* Documented average low back pain intensity of at least 6 out of 10 and greater or equal than average leg pain intensity over 7 days during screening (Numerical Rating Scale)
* Stable daily pain-related medication prescription and intake of ≤100mg morphine-equivalents
* Capacity to describe and rate pain intensity, complete study measurements, and use the study device (e.g. patient remote control, charger, diary ratings) (physician discretion)

Key Exclusion Criteria:

* Presence of pain or psychological condition that in the opinion of the investigator may interfere with the subject's ability to rate their pain and communicate such ratings
* Previous Spinal Cord Stimulation trial or is already implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Eldabe, MD, Principal Investigator — James Cook University Hospital
Locations (2):
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - James Cook University Hospital, Middlesbrough

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 subjects were enrolled in the study. 10 were withdrawn prior to randomization. 6 were randomized. Statistically relevant conclusions cannot be made from this small sample size.
Groups:
- Alternative Then Bipolar Field Shape Stimulation: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System: Spinal cord stimulation for the management of chronic neuropathic pain programmed with alternative field stimulation for 21 days, then bipolar shape stimulation for 21 days
Period: First Intervention, 21 Days
Arm/Group | Bipolar Then Alternative Field Shape Stimulation | Alternative Then Bipolar Field Shape Stimulation
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0
Period: Second Intervention, 21 Days
Arm/Group | Bipolar Then Alternative Field Shape Stimulation | Alternative Then Bipolar Field Shape Stimulation
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bipolar Then Alternative Field Shape Stimulation | Alternative Then Bipolar Field Shape Stimulation | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Patient Preferred Field Shape
Description: Number of participants preferring bipolar field shape and alternative field shape
Time Frame: 42 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Bipolar Then Alternative Field Shape Stimulation | Alternative Then Bipolar Field Shape Stimulation
Number analyzed (Participants) | 2 | 4
Participants
  Preferred Bipolar Field Shape | 2 | 2
  Preferred Alternative Field Shape | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events reported from randomization to 42 days post randomization
Groups:
- Bipolar Field Shape Stimulation: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System: Spinal cord stimulation for the management of chronic neuropathic pain programmed with bipolar field shape stimulation for 21 days
- Alternative Field Shape Stimulation: Boston Scientific's Precision SPECTRA™ Spinal Cord Stimulation System: Spinal cord stimulation for the management of chronic neuropathic pain programmed with alternative field shape stimulation for 21 days
Arm/Group | Bipolar Field Shape Stimulation | Alternative Field Shape Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02916498/Prot_000.pdf